CLINICAL TRIAL: NCT04975204
Title: A Phase I Clinical Trial Evaluating the Tolerance and Pharmacokinetics of TQB3909 Tablets in Patients With Relapsed or Refractory Advanced Malignant Tumors
Brief Title: A Clinical Trial of TQB3909 Tablets in Subjects With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3909-I-01
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3909 Tablets (Experimental): Take 100-1200mg once a day; Oral administration on an empty stomach, 28 days as a cycle.
  Interventions: Drug: TQB3909 Tablets

INTERVENTIONS:
Drug: TQB3909 Tablets — TQB3909 is an inhibitor targeting BCL-2 protein

SUMMARY:
TQB3909 is an inhibitor targeting at B-cell lymphoma (BCL)-2 protein. By binding to BCL-2 protein, TQB3909 releases Pro apoptotic proteins such as BCL-2-Anatagonist/Killer 1(BAK), BCL-2 associated X (BAX) protein and BCL-2 associated death (BAD) protein, promotes the release of cytochrome c from mitochondria, phosphatidylserine eversion, stimulates caspase 3 / 7 activity and caspase 3 / 9 cleavage, and induces apoptosis.

ELIGIBILITY:
Inclusion Criteria:

* The subjects volunteered to join the study and signed informed consent form (ICF)with good compliance.
* Age: ≥ 18 years old (when signing ICF); Eastern Cooperative Oncology Group (ECOG) performance status score: 0-1; The expected survival period is more than 3 months.
* Advanced malignant tumor diagnosed by histology or cytology.
* Relapse or failure after previous standard treatment, or intolerance to standard treatment, and no other better treatment options.
* Subject population:a)Dose escalation stage: non-Hodgkin's lymphoma;b) Dose expansion stage: non-Hodgkin's lymphoma, plasmacytoma, acute myeloid leukemia, myelodysplastic syndrome, etc.
* At least 1 lesion / measurable disease for efficacy evaluation.
* The function of main organs are well, and the following examination results are good: routine blood examination, biochemical examination, blood coagulation function examination, and heart color Doppler ultrasound evaluation.
* Female subjects of childbearing age should agree to use contraceptive measures (such as intrauterine device, contraceptive or condom) during the study period and within 6 months after the end of the study; The serum pregnancy test iss negative within 7 days before the enrollment and must be non-lactating subjects; Male subjects should agree to avoid childbirth during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Combined disease and History:

  1. There were other malignant tumors in 3 years before the first medication. The following two cases can be included: other malignant tumors treated by single operation have achieved 5-year disease-free survival (DFS) in a row; The cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non-invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  2. The diagnosis was Burkitt lymphoma, lymphoblastic lymphoma / leukemia, etc;
  3. Central nervous system (CNS) invasion was found;
  4. He has received allogeneic hematopoietic stem cell transplantation in the past;
  5. Autologous hematopoietic stem cell transplantation was performed 3 months before the first administration;
  6. There are many factors influencing oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
  7. Unrelieved toxicity of ≥ circulating tumor cells(CTC) AE 1 due to any previous treatment, excluding alopecia;
  8. Major surgical treatment, open biopsy and obvious traumatic injury were performed within 28 days before the study;
  9. There are active or uncontrolled primary autoimmune hemocytopenia, including autoimmune hemolytic anemia (AIHA), idiopathic thrombocytopenic purpura (ITP), etc;
  10. Arteriovenous thrombotic events occurred within 6 months before the first medication, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
  11. Have a history of psychotropic drug abuse and can not quit or have mental disorders;
  12. Subjects with any severe and / or uncontrolled disease included:

      1. Patients with ≥ 2 grade myocardial ischemia 6 months between the first administration or myocardial infarction, arrhythmia (male corrected QT interval (QTc) > 450ms, female QTc > 470ms) and ≥ 2 grade congestive heart failure (NYHA classification), Cardiac color Doppler ultrasound to evaluate left ventricular ejection fraction（LVEF）<50%;
      2. There was active severe infection (≥ CTC AE grade 2 infection);
      3. Fever and neutropenia were found within 1 week before the first medication;
      4. Diabetes was poorly controlled (fasting blood glucose (FBG) > 10mmol/L).
      5. Active hepatitis *;

         * active hepatitis (hepatitis B reference: hepatitis B surface antigen (HBsAg) positive, and hepatitis B virus(HBV) DNA detection value > 2000 copies /mL or 500 internation unit (IU)/mL; Hepatitis C reference: hepatitis C virus(HCV) antibody was positive, and HCV titer detection value exceeded the upper limit of normal value);
      6. History of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or organ transplantation;
      7. Patients with epilepsy and need treatment.
* tumor related symptoms and treatment:

  1. Subjects who have received chemotherapy, radiotherapy within 4 weeks prior to the first dose or received immune checkpoint inhibitors and CAR-T treatment 12 weeks before the first medication, or other anti-tumor treatment within 5 half-life prior to the first dose (the washing and removing period is calculated from the end of the last treatment) ;
  2. Subjects who have previously received BCL-2 inhibitors.
* Subjects who have received the vaccine within 4 weeks prior to the first dose, or is planning to be vaccinated during the study period.
* Subjects who have participated in clinical trials of other anti-tumor drugs within 4 weeks before the first dose.
* According to the judgment of the investigator, subjects with concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects with other reasons which are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | up to 18 months
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Recommended Phase II Dose (RP2D) | up to 18 months
  DLT describes side effects of a drug or other treatment that are serious enough to To evaluate RP2D of TQB3909 tablets in adult patients with advanced solid tumors

SECONDARY OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) | up to 18 months
  The incidence and severity of AEs and SAEs, as well as abnormal laboratory test indicators.
Time to reach maximum(peak )plasma concentration following drug administration (Tmax) | Within 32 weeks after administration
  To characterize the pharmacokinetics of TQB3909 by assessment of time to reach maximum plasma concentration after single and multiple dosing
Maximum (peak) plasma drug concentration (Cmax) | Within 24 hours after administration
  Cmax is the maximum plasma concentration of TQB3909.
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Css-max) | Within 32 weeks after administration
  Css-max is the steady state maximum concentration of TQB3909 .
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | Within 24 hours after administration
  To characterize the pharmacokinetics of TQB3909 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Area under the plasma concentration-time curve from time zero to infinity(AUC0-∞) | Within 24 hours after administration
  To characterize the pharmacokinetics of TQB3909 by assessment of area under the plasma concentration time curve from the first dose to infinity.
Area under the plasma concentration-time curve when reaching steady state (AUCss) | Within 32 weeks after administration
  AUCss is the area under the curve of TQB3909.
Apparent total clearance of the drug from plasma after oral administration (CL/F) | Within 24 hours after administration
  CL/F is total clearance rate for TQB3909.
Elimination half-life (t1/2) | Within 24 hours after administration
  t1/2 is time it takes for the blood concentration of TQB3909 to drop by half.
Mean residence time (MRT) | Within 24 hours after administration
  MRT describes the average time that TQB3909 remains in the body.
Minimum steady-state plasma drug concentration during a dosage interval (Css-min) | Within 32 weeks after administration
  Css-min is the minimum plasma concentration of TQB3909.
Degree of fluctuation(DF) | Within 32 weeks after administration
  DF is the volatility coefficient of TQB3909.
Average steady-state plasma drug concentration during multiple-dose administration (Css-av) | Within 32 weeks after administration
  Css-av is the average of steady-state plasma concentration of TQB3909 .
Apparent volume of distribution after non-intervenous administration (Vd/F) | Within 24 hours after administration
  Vd/F is the bioavailability corrected apparent distribution volume of TQB3909
Progression-free survival (PFS) | up to 18 months
  PFS is defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall response rate (ORR) | up to 18 months
  Percentage of participants achieving complete response (CR) and partial response (PR).
Complete response rate（CRR） | up to 18 months
  CRR refers to the percentage of patients who enter the clinical disappearance period of the disease after a certain treatment.
Disease control rate（DCR） | up to 18 months
  Percentage of participants achieving CR and PR and stable disease (SD).
Duration of Response (DOR) | up to 18 months
  The period from the participants first achieving CR or PR to disease progression.
Overall survival (OS) | up to 18 months
  OS is defined as the time from the first administration to all-cause death.
Protein concentration or gene expression level related to BCL-2 signaling pathway | up to 18 months
  To evaluate the changes of BCL-2 signaling pathway related to proteins or genes.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Institute of Hematology & Blood Diseases Hospital,Chinese Academy of Medical Sciences &Peking Union Medical College, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No